CLINICAL TRIAL: NCT00300872
Title: A Randomized, Placebo-controlled Study of the Medium-term Effect of Nasal CPAP on 24 Hour Blood Pressure and Vascular Endothelial Growth Factor in Obstructive Sleep Apnea Syndrome
Brief Title: Effect of Nasal Continuous Positive Airway Pressure (CPAP) Blood Pressure and Vascular Endothelial Growth Factor in Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Prof, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Resp/hui/2006/002
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Continuous positive airway pressure (CPAP)
  Interventions: Device: Continuous positive airway pressure (CPAP)
- 2 (Sham Comparator): Sham Continuous positive airway pressure (CPAP)
  Interventions: Device: Sham Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Continuous positive airway pressure (CPAP) - Horizon LT 8001 Continuous positive airway pressure (CPAP) device.
  Arms: 1
Device: Sham Continuous positive airway pressure (CPAP) — Sham Continuous positive airway pressure (CPAP) - Continuous positive airway pressure (CPAP) units set to the lowest pressure (4 cm of water pressure) and 6 extra 4mm holes will be inserted in the collar of the main tubing at the end of the mask to allow air escape and to prevent carbon dioxide rebreathing.
  Arms: 2

SUMMARY:
Sleep-disordered breathing (SDB) briefly means cessation of breathing during sleep at least 5 times per hour. SDB is a common disorder affecting 9 to 24% of the middle-aged and overall 4% of the middle-aged male population suffers from the Obstructive sleep apnea syndrome (OSA) i.e. Sleep-disordered breathing (SDB) with associated daytime sleepiness. Several major epidemiological studies have shown that SDB is not only an independent risk factor for hypertension but it is also strongly associated with heart failure and stroke. The mechanism for the linkage between SDB and cardiovascular consequences is not fully determined. Vascular endothelial growth factor (VEGF) is a soluble 34-46 kD angiogenic heparin-binding glycoprotein. This cytokine regulates multiple endothelial cell functions including vascular permeability and vascular tone and some data suggest that it may contribute to the atherosclerotic process. Recent studies have shown increased plasma and serum concentrations of Vascular endothelial growth factor (VEGF) in patients with OSA and there were correlations between VEGF concentrations and the severity of OSA, as indexed by the minimum oxygen saturation level and the frequency of the upper airway obstruction per hour of sleep. A recent non-randomized study with a small sample size has shown a significant decrease in Vascular endothelial growth factor (VEGF) concentrations in patients in whom nocturnal hypoxia improved after 1 year of nasal continuous positive airway pressure (CPAP) therapy.

Despite robust evidence showing improvement of symptoms, cognitive function and quality of life in obstructive sleep apnea (OSA) patients treated with nasal CPAP, there are nevertheless conflicting data whether Continuous positive airway pressure (CPAP) can reduce daytime blood pressure (BP) in patients with OSA. Two randomized placebo controlled studies have shown reduction of 24-hr systolic and diastolic blood pressure (BP) in obstructive sleep apnea (OSA) patients after 1 month of nasal continuous positive airway pressure (CPAP) therapy while other investigators have shown no such benefit.

This randomized, sham-placebo controlled study aims to assess 1) the effect of nasal continuous positive airway pressure (CPAP) over a period of 3 months on 24 hr blood pressure (BP); and 2) whether any change in BP and plasma Vascular endothelial growth factor (VEGF) is related to the baseline severity of obstructive sleep apnea (OSA) and continuous positive airway pressure (CPAP) compliance.

DETAILED DESCRIPTION:
Subjects and Methods:

We propose to carry out a prospective, randomized sham placebo-controlled parallel study on 140 consecutive patients newly diagnosed with OSA, as defined by overnight sleep study showing apnea hypopnea index (AHI) >10 per hour of sleep plus excessive daytime sleepiness or two of the following symptoms: choking or gasping during sleep, recurrent awakenings from sleep, unrefreshed sleep, daytime fatigue and impaired concentration.1 The patients will be recruited from the Respiratory Clinic, Prince of Wales Hospital, Shatin, HK.

Sleep assessment:

Overnight diagnostic polysomnography (PSG) [Healthdyne Alice 4, USA] will be performed for every subject on the first night recording electroencephalogram, electro-oculogram, submental electromyogram, bilateral anterior tibial electromyogram, electrocardiogram, chest and abdominal wall movement by inductance plethysmography, airflow measured by a nasal pressure transducer [PTAF2, Pro-Tech, Woodinville, WA, USA]and supplemented by an oral thermister, and finger pulse oximetry as in our previous studies.2-4 Sleep stages will be scored according to standard criteria by Rechtshaffen and Kales. 5 Apnoea is defined as cessation of airflow for > 10 seconds and hypopnea as a reduction of airflow of >50% for > 10 seconds plus an oxygen desaturation of > 3% or an arousal.

Following confirmation of significant obstructive sleep apnea syndrome (OSA) from the overnight sleep study with apnea hypopnea index (AHI) >10/hr, each patient will be interviewed by the physician on duty and randomized into 2 groups receiving either nasal therapeutic continuous positive airway pressure (CPAP) treatment or sham continuous positive airway pressure (CPAP), via a balanced block design, after completion of recording of 24 hr ambulatory blood pressure (BP).

Ambulatory Blood Pressure Monitoring(ABPM):

All patients with obstructive sleep apnea (OSA) will be fitted with the Ultralite Ambulatory Blood Pressure Monitoring (ABPM) (Spacelabs Medical, Redmond, WA) via an arm cuff as out-patients during normal activities and monitored for 48 hrs prior to commencement of therapeutic or sham continuous positive airway pressure (CPAP) treatment. The patients' arm circumference will be measured at the biceps level and an appropriate sized arm cuff will be applied. The machine will be programmed for cuff inflation measurement every 30 minutes for 48 hrs and can only be removed for bathing. Patients will be asked to abstain from caffeine-containing products during this time but to continue their normal daily activities. Patients will record the time they retire to bed and the subsequent time of waking in order to identify the sleep period. Data gathered before 6pm on the second evening will be discarded to allow for acclimatization and the analysis will be performed with the second 24 hr of data (6pm to 6am).6 Data will be manually checked for artifact by our respiratory fellow, who will be blinded to the treatment status of the patient. Forty-eight hrs before the end of the therapeutic or sham continuous positive airway pressure (CPAP) at 3 months, the patients will be fitted with the Ambulatory Blood Pressure Monitoring(ABPM) machine and the same procedure repeated.

Measurement of blood samples:

Fifteen ml of fasting venous blood will be taken from each patient after the overnight PSG. Plasma will be separated within 2 hours in a refrigerated centrifuge, aliquoted and stored at -70C until assayed. Plasma VEGF will be measured by a quantitative enzyme-linked immunoassay technique using a commercially available kit (R & D Systems, Abingdon, UK). Serum lipids will be checked as it has been reported that Vascular endothelial growth factor (VEGF) also increases in patients with hyperlipidemia, with and without atherosclerosis.7

Therapeutic continuous positive airway pressure (CPAP) vs Sham placebo:

Patients in the therapeutic continuous positive airway pressure (CPAP) or sham continuous positive airway pressure (CPAP) treatment arm will be offered a 30-minute daytime trial of nasal continuous positive airway pressure (CPAP) treatment. Each patient will be given a basic continuous positive airway pressure (CPAP) education program by our respiratory nurse supplemented by education brochure.4 The nurse will fit a comfortable continuous positive airway pressure (CPAP) mask from a wide range of selection for the patient, who will then be given a short trial of continuous positive airway pressure (CPAP) therapy with the Autoset (Resmed, Sydney, Australia) continuous positive airway pressure (CPAP) device for those in the therapeutic continuous positive airway pressure (CPAP) arm for approximately 30 minutes for acclimatization in the afternoon. Attended continuous positive airway pressure (CPAP) titration will be performed with the Autoset auto-titrating device on the second night of the PSG study for the group randomized to the therapeutic continuous positive airway pressure (CPAP) arm.2-4 All the patients in the therapeutic continuous positive airway pressure (CPAP) arm will be prescribed the Horizon LT 8001 continuous positive airway pressure (CPAP) device (De Vilbiss, Somerset, PA, USA) with a time counter recording machine run time. The continuous positive airway pressure (CPAP) pressure for each patient will be set at the minimum pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night as determined by the overnight Autoset continuous positive airway pressure (CPAP) titration study.

The patients randomized to the subtherapeutic continuous positive airway pressure (CPAP) arm will have the CPAP units set to the lowest pressure (4 cm of water pressure) and 6 extra 4mm holes will be inserted in the collar of the main tubing at the end of the mask to allow air escape and to prevent carbon dioxide rebreathing.8,9 They will be given a trial of 30 minutes for acclimatization before starting continuous positive airway pressure (CPAP) at home.

All the patients in each arm will be followed up at the Respiratory clinic separately at 1 month and 3 months and the objective continuous positive airway pressure (CPAP) compliance will be measured from the time counter. Although the 2 different treatment arms are explained in the patient information, the patients will not be aware of whether they are receiving therapeutic or sham continuous positive airway pressure (CPAP). The research nurse responsible for randomization of patients to different treatment arms will not participate in outcome assessments, which will be conducted by a different team of nurses who are not aware of the randomization status of the patients.9 At the end of the study (ie 3 months), all patients in the subtherapeutic continuous positive airway pressure (CPAP) arm will be readmitted for AutoSet continuous positive airway pressure (CPAP) titration to establish their long-term therapeutic pressure.

Other outcome assessment:

Prior to commencement of nasal therapeutic or sham continuous positive airway pressure (CPAP), all patients have to go through several measurements. These include assessment of subjective sleepiness with the Epworth sleepiness scale (ESS)10, quality of life with the Calgary Sleep Apnea Quality of Life Index (SAQLI).11 The ESS is a questionnaire specific to symptoms of daytime sleepiness and the patients are asked to score the likelihood of falling asleep in eight different situations with different levels of stimulation, adding up to a total score of 0 to 24.10 The Calgary Sleep Apnea Quality of Life Index (SAQLI) has 35 questions organized into four domains: daily functioning, social interactions, emotional functioning and symptoms with a fifth domain, treatment-related symptoms, to record the possible negative impacts of treatment. The Sleep Apnea Quality of Life Index (SAQLI) has a high degree of internal consistency, face validity as judged by content experts and patients and construct validity as shown by its positive correlations with the Short Form-36 Health Survey questionnaire (SF-36) and the improvement in scores in patients successfully completing a 4 weeks' trial of continuous positive airway pressure (CPAP).11 It contains items shown to be important to patients with sleep apnea and is designed as a measure of outcome in clinical trials in sleep apnea, and has been applied previously in our Chinese obstructive sleep apnea (OSA) patients on continuous positive airway pressure (CPAP). 4 All patients will have to complete the Epworth Sleepiness Score (ESS) and Sleep Apnea Quality of Life Index (SAQLI) at baseline, 1 month and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80 yrs
* Apnea hypopnea index (AHI) > 10/hr on Polysomnograph (PSG) with symptoms of obstructive sleep apnea (OSA) as described previously
* Epworth Sleepiness Scale (ESS) >10
* Patients with hypertension will still be eligible to enter and continue the study as long as there is no alteration of anti-hypertensive medications during the study period

Exclusion Criteria:

* Patients having problems staying awake during driving, shift work
* Recent myocardial infarction
* Unstable angina
* Underlying malignancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2005-01; Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Change in 24 hr mean blood pressure at 3 months | baseline and 3 months

SECONDARY OUTCOMES:
Changes in systolic and diastolic blood pressure, changes in mean blood pressure awake and asleep, change in plasma Vascular endothelia growth factor (VEGF) at 3 months | baseline and 3 months
Whether any change in blood pressure or vascular endothelial growth factor (VEGF) is related to the baseline severity of obstructive sleep apnea (OSA) and continuous positive airway pressure (CPAP) compliance over 3 months | baseline and 3 months
Epworth Sleepiness Scale (ESS) and Calgary Sleep Apnea Quality of Life Index (SAQLI) at 1 month and 3 months. | baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong